CLINICAL TRIAL: NCT01162395
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD3514 in Patients With Metastatic Castration-Resistant Prostate Cancer.
Brief Title: Open Label Prostate Cancer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3760C00001; 2010-020232-19 (EudraCT Number); IND 111707
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Tumour; Castration Resistant; Prostate Androgen Receptor Down Regulator; Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — AZD3514

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Ascending doses of AZD3514 administered orally to patients to define the maximum tolerated dose (MTD)
  Interventions: Drug: AZD3514

INTERVENTIONS:
Drug: AZD3514 — Patients will be given AZD3514 orally as a single dose, and then multiple once daily dosing following a 5-9 day washout.

SUMMARY:
The main purpose of the study is to investigate the safety and tolerability of AZD3514 when given orally to patients with castration-resistant prostate cancer (CRPC)

ELIGIBILITY:
Inclusion Criteria:

* Males aged 20 years or older.
* Histologically or Cytologically proven diagnosis of prostate cancer for which no standard therapy is currently considered appropriate.
* Documented evidence of metastatic prostate cancer
* Presence of progressive disease defined as one or more:
* Biochemical progression of the prostate cancer
* Progression as defined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 guidelines
* Two or more new metastatic bone lesions from bone scans from a previous assessment
* Serum testosterone concentration less or equals 50 ng/dL
* World Health Organization (WHO) performance status 0 to 1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.
* Sexually active males should be willing to use condoms
* For inclusion in the AZD3514 administered in combination with abiraterone acetate cohort(s), patients must:
* Have received prior chemotherapy containing or based on docetaxel
* Not have received prior treatment with abiraterone acetate, MDV3100, TAK700, TOK001 or other similar therapies which target the AR axis or with selective AR down-regulator-like properties
* For inclusion in the AZD3514 administered in combination with abiraterone acetate in patients who are currently receiving abiraterone acetate cohort(s), patients must:

  1. Have been stable on abiraterone acetate abiraterone acetate for ≥ 4 months (i.e. stable PSA values) and have achieved ≥ 50% reduction in PSA while being treated with abiraterone acetate
  2. Have evidence of biochemical progression (PSA) of the prostate cancer, as defined in inclusion number 5 (except for the withdrawal of abiraterone acetate as an anti-androgen therapy)
* For inclusion in the paired (same lesion) tumour biopsy research, patients must:

  1. Provide informed consent for paired tumour biopsy sampling
  2. Have bone or soft tissue lesions that are suitable for paired biopsy sampling

Exclusion Criteria:

* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAEv4) grade 1 except for alopecia or toxicities related to the use of gonadotropin-releasing hormone agonists
* Medically important spinal cord compression or brain metastases
* Medically important evidence of severe or uncontrolled systemic disease
* History of hypersensitivity to active or inactive excipients of AZD3514 or drugs with a similar chemical structure or class to AZD3514
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD3514
* Inadequate bone marrow reserve or organ function
* Any medically important factors identified from electrocardiogram (ECG) measurements
* Concurrent or recent treatment with certain medications or medical procedures

The following criteria exclude patients from entering the AZD3514 administered in combination with abiraterone acetate cohort(s):

* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases or conditions, including adrenocortical insufficiency or a history of cardiovascular disease including heart failure (currently there are no randomized data for the use of abiraterone acetate in patients with LVEF < 50% or NYHA Class III or IV heart failure), which would make it undesirable for the patient to participate in the trial. See the full local prescribing information for abiraterone acetate for more detail
* Child-Pugh class B and C hepatic impairment
* If unable to fast for ≥ 2 hours prior to taking a dose to ≥ 1 hour post dose
* Received abiraterone acetate treatment previously
* Known hypersensitivity to components of prednisone or prednisolone
* Any systemic fungal infections

Ages: 20 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of AZD3514 when given orally to patients with CRPC. | At every visit.

SECONDARY OUTCOMES:
To define the MTD, if possible, a lower biologically-effective dose(s) or maximum feasible dose (if decided by the Safety Review Committee (SRC) and AstraZeneca). | After each Cohort.
To characterise the PK of AZD3514 after a single oral dose and at steady state after multiple oral doses. | After each Cohort.
To obtain an assessment of the activity of AZD3514 as monotherapy and/or in combination with abiraterone acetate on the circulating levels of prostate-specific antigen (PSA). | Visits 1, 4, 6, 7, 9, 10, follow-up visits, discontinuation visit
To obtain a preliminary assessment of the anti-tumour activity of AZD3514 as monotherapy and/or in combination with abiraterone acetate by evaluation of counts of Circulating Tumour Cells (CTCs). | Visits 1, 6, 8, 9, 10, follow-up visits, discontinuation visit
To obtain an assessment of the activity of AZD3514 as monotherapy and/or in combination with abiraterone acetate on the circulating levels of prostate-specific antigen (PSA). | Visits 1, 10, follow-up visits, discontinuation visit
To investigate safety, tolerability, MTD (and/or biologically-effective dose(s) or maximum feasible dose) and PK of AZD3514 and abiraterone when administered in combination, in patients who have not received prior treatment with abiraterone acetate | At every visit
To compare the PK of AZD3514 monotherapy in patients who have been fed or fasted before the administration of study treatment | At visits 2 and 4
To investigate the effect of AZD3514 on biomarkers of AR expression in paired pre- and post-dose tumour biopsies. | July 2012 - Feb 2013

CONTACTS AND LOCATIONS:
Overall Officials: Tony Elliott, MD, Principal Investigator — The Christie Hospital; Glen Clack, MD, Study Director — AstraZeneca
Locations (5):
- Research Site, Portland, Oregon, United States
- Research Site, Amsterdam, Netherlands
- United Kingdom (3):
  - Research Site, Glasgow
  - Research Site, Manchester
  - Research Site, Surrey

REFERENCES:
- [Derived] James GD, Symeonides SN, Marshall J, Young J, Clack G. Continual reassessment method for dose escalation clinical trials in oncology: a comparison of prior skeleton approaches using AZD3514 data. BMC Cancer. 2016 Aug 31;16(1):703. doi: 10.1186/s12885-016-2702-6. PMID 27581751
- See also: D3760C00001 Clinical Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1380&filename=D3760C00001_Clinical_Trial_Disclosure_Synopsis.pdf